CLINICAL TRIAL: NCT02868398
Title: Efficacy and Safety of Golimumab in Maintaining Deep Remission and Quality of Life in Ulcerative Colitis Patients in Deep Prolonged Remission With Infliximab. An Open Label, Non Interventional One Year Study.
Brief Title: Efficacy of Golimumab in Maintaining Deep Remission in UC Patients in Prolonged Remission With Infliximab
Acronym: Switch
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Director gastroenterologist, Evangelismos Hospital
Other Study IDs: 143/27-06-2016
Record Dates: First submitted 2016-07-07; First posted 2016-08-16 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Golimumab; Deep and prolonged remission
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study monitors the efficacy and safety of Golimumab in maintaining deep remission and quality of life in Ulcerative Colitis patients in deep prolonged remission with Infliximab. Patients will be followed up for one year and they will be assessed with biochemical tests (C-Reactive Protein , Full Blood Count , Faecal Calprotectin),endoscopic evaluation (MAYO Score) and finally histologically.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic idiopathic relapsing-remitting or continuously active inflammatory bowel disease (IBD) which almost exclusively affects the colonic mucosa. Acute severe flares of UC may lead onto potential lethal complications, such as massive haemorrhage, toxic megacolon, peritonitis, and colectomy whereas chronic active disease may lead to functional failure of the large bowel, dysplasia and colorectal cancer. Traditional therapeutic targets, such as normalization of stools and absence of rectal bleeding, are no longer considered sufficient to prevent the aforementioned long term sequelae of uncontrolled colonic inflammation. Thus, new therapeutic targets are emerging which aim at achieving optimal long-term outcomes of UC. Along this line, therapy is moving from mere control of symptoms towards a more global control of inflammation by achieving and maintaining long-term complete clinical remission (relief of abdominal pain, normalization of stools, and cessation of rectal bleeding), normalization of serologic (white blood cells and C-Reacting Protein) and faecal markers of inflammation (calprotectin), and endoscopic (normal looking mucosa) and histologic remission (absence of acute and chronic inflammation on biopsies from the affected colonic areas). This composite definition of remission (namely 'complete' or 'deep' remission) consisting of appropriate patient reported outcomes (PROs) and objective markers of intestinal inflammation may be associated with improved long-term outcomes of disease, such prevention of complications, hospitalizations, and colectomy, avoidance of disability and maintenance of at least near-normal patient quality of life. This composite clinical and biological remission along with mucosal healing and histologic remission is now considered as a realistic therapeutic goal.

Patients fulfilling the inclusion criteria and willing to participate will receive golimumab therapy subcutaneously for 1 year.

Patients will be followed in the outpatient IBD Clinic at 3-month intervals as is the usual practice in our department. At each visit patients will undergo clinical evaluation using the Partial Mayo score, physical examination, monitor of body weight and body mass index, and routine laboratory tests which are included in routine clinical practice of treatment with biologic agents in IBD (FBC, Estimated Sedimentation Rate, CRP, Liver Function Tests, Urea, Creatinine, serum glucose and electrolytes, and faecal calprotectin) in order to ensure effectiveness and safety of treatment. In each visit, patients will fill questionnaires to assess quality of life, disability, work productivity, and satisfaction with therapy. The daily bowel frequency, rectal bleeding, presence and grading of abdominal pain and the overall subjective condition of patient's general health between visits will be recorded daily in pre-administered diaries.

After 1 year of golimumab administration patients will be re-evaluated by endoscopy and biopsies in order to define the percentage of patients that remain at deep remission.

For those patients presenting with a flare of disease during the 1 year follow up, treatment will be individualized depending on the severity of the flare.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA
* Clinical remission as assessed by PROs 1 and 2 of the Mayo score
* Biochemical remission, as assessed by a normal full blood count, erythrocyte sedimentation rate, C-Reacting Protein, and faecal calprotectin,
* Endoscopic remission, defined as an endoscopic subscore of the Mayo score equal to 0 or 1.
* Written informed consent.

Exclusion Criteria:

* Flare up of Ulcerative Colitis.
* Non endoscopic remission.
* Co-administration of Immunosuppressive drugs or/and topical use of Mesalazine.
* Allergic reaction to Infliximab or previously Infliximab dose over 5mg/Kg/8 weeks.
* Infection during study.
* Consent form not signed by the patient.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ulcerative colitis patients in deep remission after 2 years of infliximab administration
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of golimumab in maintaining deep remission with patients with UC. Patient will complete the short Inflammatory Bowel Disease Questionnaire (short SIBDQ) and Treatment Satisfaction Questionnaire for Medication (TSQM) form. | 1 year
  The primary outcome will be to assess the efficacy o Golimumab to maintain deep remission of UC

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Viazis, Director, Principal Investigator — Evangelismos Hospital
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided